CLINICAL TRIAL: NCT05947877
Title: Effectiveness of Interventional Non-Pharmacological Nursing Pain Management for Preterm Infants at Neonatal Intensive Care Unit
Brief Title: Non-Pharmacological Nursing Pain Management for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Collaborators: Numan Nafie Hameed (Unknown)
Responsible Party: Principal Investigator, Hiba Abdulwahid Dawood, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Preterm Infant Pain Management
Record Dates: First submitted 2023-06-29; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Pain Management
Keywords: Non-pharmacological Pain Management Strategies; Preterm Infants; NICU
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Preterm infants and their mothers were masked from the nature of the administered intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Non-pharmacological nursing pain management strategies (Experimental): This arm considers conventional care.
  Interventions: Procedure: Non-pharmacological pain management strategies
- Breast milk (Experimental): This arm considers breast milk. The preterm infants were orally fed 2 ml of expressed breast milk through a syringe 2 minutes before heel stick over the anterior surface of the tongue, allowing for preterm infant swallowing rates over a period of 1-2 minutes. Thereafter, the bedside nurse conducts the heel lancing. When the mother is present with her preterm infant in the NICU, the breast milk was expressed by the mother and provided in a syringe at least 30 minutes before the intervention (n = 11). For the rest 10 preterm infants whose mothers were not present with them in the NICU, they send their breast milk to be kept in the NICU refrigerator. This milk was first warmed in room temperature 30 minutes before it was given to the preterm infant.
  Interventions: Procedure: Non-pharmacological pain management strategies
- Oral sucrose (Experimental): This arm considers oral sucrose. The researchers gave one ml of 24% oral sucrose to the preterm infant two minutes prior to the heel stick, drop-by-drop via syringe over the anterior surface of the tongue which enable the preterm infant to swallow rates over a period of 1-2 minutes. Conducting the heel stick procedure with lancet approximately two minutes after administering the sucrose. The pharmacy at the study site supplies the syringes containing the oral sucrose solution, solutions are prepared and packaged in an identical matter, the SR will label each syringe with the preterm infants' study number and name to ensure added protection.
  Interventions: Procedure: Non-pharmacological pain management strategies
- KMC (Experimental): This arm considers KMC. The preterm infants were randomized to the KMC intervention; the researchers explained to the mother that she and her preterm infants will be put in KMC position, where the diaper-clad infant was held upright, at an angle of approximately 60°, between the mothers' breasts, providing maximal skin-to-skin contact between mother and baby. A blanket was placed over the preterm infant's back, and the mother's clothes were wrapped around the neonate, the preterm infant will remain in KMC for 30 minutes before the lancing procedure, during, and at least 30 minutes after the heel lance.
  Interventions: Procedure: Non-pharmacological pain management strategies
- Nesting position (Experimental): This arm considers nesting position. Before heel lancing, the researchers prepared and arranged all the required nesting equipment from the NICU such as linen, small pillow, and blanket. Making the nest by folding the blanket form one corner, then placing it upright and laying the linen over the blanket. Positioning the preterm infant inside the nest in supine position, ensuring that the nest size is suitable for the preterm infant's body, neither too loose nor too tight during nesting position. Position the preterm infant first in supine position through wrapping infant with hand to midline the nest through putting small pillow under the preterm infant's shoulder to keep airway open, the nested infants were placed in nest, that helped to maintain and support them in a flexed position but still facilitated unrestricted movement of their body and limbs, supine nesting position conducting 30 minutes before heel lancing and, during, and after the procedure for 30 minutes.
  Interventions: Procedure: Non-pharmacological pain management strategies

INTERVENTIONS:
Procedure: Non-pharmacological pain management strategies — Non-pharmacological pain management strategies

SUMMARY:
A randomized controlled trial will be conducted to examine the effect of non-pharmacological nursing pain management strategies in alleviating pain among preterm infants. The study includes a simple random sample of 105 preterm infants with CGA 32- < 37 weeks were randomly assigned into five groups: routine care (n = 21), breast milk (n = 21), oral sucrose (n = 21), KMC (n = 21), nesting position (n = 21). PIPP-R will be used to subjectively assess the pain intensity after heel stick, and salivary cortisol measures will be used to objectively assess the pain intensity in NICU at Children Welfare Teaching Hospital/ Medical City Complex in Baghdad City.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants whose corrected gestational age from (32 - <37) weeks of pregnancy,
* Preterm infants who do not experience any painful procedure for last 24 hours.
* Preterm infants who do not receive any sedation for last 24 hours, and clinically required heel stick.

Exclusion Criteria:

* Full-term infants whose gestational age (GA) is >37 weeks
* Preterm infants who extremely preterm (< 28 weeks); very preterm (28-< 32 weeks)
* Preterm infants who are proven or suspected sepsis, major congenital malformations, heart defect, necrotizing enterocolitis (NEC), and neurodevelopmental disability.
* Preterm infants who receive respiratory support {Mechanical Ventilation, Continuous Positive Airway Pressure (CPAP), or high-flow support}
* Preterm infants who are indicated for surgery
* Preterm infants who are contraindicated to oral sucrose
* Twins
* Preterm infants who had a condition that might influence their physiological and responses to pain, e.g., congenital anomalies or severe illnesses requiring treatment with antiepileptics, muscle relaxants, or analgesic drugs.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile - Revised | Two months
  Premature Infant Pain Profile - Revised measures pain intensity through infant indicators (heart rate, oxygen saturation, brow bulge, eye squeeze). Other indicators in the PIPP-R include gestational age and behavioral state.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Nursing- The University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided